CLINICAL TRIAL: NCT04160091
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of FX006 in Patients With Glenohumeral Osteoarthritis or Shoulder Adhesive Capsulitis (RANGE)
Brief Title: Study to Evaluate the Efficacy and Safety of FX006 in Patients With Glenohumeral Osteoarthritis or Shoulder Adhesive Capsulitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely due to the COVID-19 pandemic creating uncertainty impacting trial progress and costs.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX006-2018-016
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Shoulder; Adhesive Capsulitis
Keywords: Osteoarthritis; Adhesive Capsulitis; Shoulder; Pain; Intra-articular; Injection; Steroid
MeSH Terms: conditions — Bursitis; Osteoarthritis; Pain | interventions — FX006; Triamcinolone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FX006 32mg in Glenohumeral OA Population (Experimental): Single intra-articular (IA) injection
  Interventions: Drug: FX006
- Normal Saline in Glenohumeral OA Population (Placebo Comparator): Single intra-articular (IA) injection
  Interventions: Drug: Normal Saline
- FX006 32mg in Adhesive Capsulitis Population (Experimental): Single intra-articular (IA) injection
  Interventions: Drug: FX006
- Normal Saline in Adhesive Capsulitis Population (Placebo Comparator): Single intra-articular (IA) injection
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: FX006 — Single intra-articular injection
  Other Names: Zilretta
  Arms: FX006 32mg in Adhesive Capsulitis Population; FX006 32mg in Glenohumeral OA Population
Drug: Normal Saline — Single intra-articular injection
  Arms: Normal Saline in Adhesive Capsulitis Population; Normal Saline in Glenohumeral OA Population

SUMMARY:
This is a double-blind study to evaluate the efficacy and safety of FX006 in patients with glenohumeral osteoarthritis (OA) or shoulder adhesive capsulitis (AC).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group study in separate cohorts of patients with a documented history of either glenohumeral OA or shoulder AC. Glenohumeral OA and shoulder AC patients will be randomized to receive a single intra-articular injection of either FX006 or placebo (saline) in a 1:1 ratio to the index shoulder with a 24-week Treatment Evaluation Period. Glenohumeral OA patients will be stratified by Baseline average daily shoulder pain with movement score according to the following classifications: 5.0 to <7.0 or ≥7.0 to 9.0 (0 to 10 numeric rating scale [NRS]). Shoulder AC patients will be stratified by Baseline average daily shoulder pain with movement score according to the following classifications: 5.0 to <7.0 or ≥7.0 to 9.0 (0 to 10 NRS), and by pain duration since onset (1 to 3 months, inclusive, or >3 to ≤6 months). A Home Exercise Program will be implemented 3 days following injection for shoulder AC patients.

ELIGIBILITY:
Inclusion Criteria:

Glenohumeral OA:

* Male or female, 35 to 80 years of age, inclusive, on the day of consent.
* Painful symptoms associated with OA of the index glenohumeral joint for ≤3 months prior to the Screening Visit.
* Grade 2 or 3 OA in the index glenohumeral joint based on the Samilson-Prieto classification system as confirmed by X-ray (axillary view and true anterior-posterior view) taken at the Screening Visit.

Shoulder AC:

* Male or female, 35 to 80 years of age, inclusive, on the day of consent.
* Pain associated with AC of the index joint for ≥1 month but ≤ 6 months prior to the Screening Visit.
* Limitations on both active and passive ROM ≥25% in at least 2 directions (e.g., forward flexion, abduction, and internal and external rotation assessed in a standardized protocol) compared with the contralateral shoulder or with normal values.
* No X-ray evidence of OA of the index shoulder (axillary view and true anterior-posterior view) at the Screening Visit.
* Agrees to complete a standardized, protocol-specified shoulder Home Exercise Program (HEP) starting 3 days after injection until the End of Study (EOS) Visit.

Both:

* Written consent to participate in the study
* Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions
* (BMI) ≤ 40 kg/m2
* Average daily mean shoulder pain with movement score ≥5.0 and ≤9.0 in the index shoulder (0 to 10 NRS) using the average daily ratings for at least 5 out of the 7 days prior to Day 1.
* Shoulder pain present >15 days in the month prior to the Screening Visit
* Willing to complete a washout of protocol-specified excluded medications 7 days prior to Day 1 and abstain from use of protocol-specified excluded medications throughout the study
* Willing to abstain from nonpharmacological therapies for the index joint for 2 weeks prior to Day 1 and throughout the study.

Exclusion Criteria:

* Has both glenohumeral OA and shoulder AC
* Has bilateral AC
* Has bilateral glenohumeral OA with glenohumeral OA pain of the shoulder contralateral to the index shoulder >3.0 (0 to 10 NRS) within 1 month prior to the Screening Visit
* Has a history of arthritis in other joints of the index shoulder (as confirmed by medical history and physical exam)
* Has a history or suspicion of full thickness rotator cuff tear in the index shoulder within 6 months of the Screening Visit
* Has symptomatic partial rotator cuff tear, tendinopathy, tendonitis, or bursitis in the index shoulder within 6 months of the Screening Visit
* Has a subchondral bone insufficiency fracture or humeral head necrosis/collapse in the index shoulder
* Shoulder AC patients only: Has a history of shoulder surgery or radiotherapy
* Glenohumeral OA patients only: Has a previous shoulder injury with functional limitation ≥1 month or surgery within 52 weeks of the Screening Visit
* Has an index shoulder with major dysplasia or congenital abnormality, osteochondritis dissecans, acromegaly, ochronosis, hemochromatosis, Wilson's disease, or primary osteochondromatosis, or a history of avascular necrosis with secondary OA
* Has current or history of infection in the index shoulder or current skin infection at injection site
* Has a concurrent chronic pain condition with a pain score >3.0 (0 to 10 NRS) within 1 month prior to the Screening Visit
* Has a history or current evidence of reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease, systemic lupus erythematosus, calcium pyrophosphate dihydrate crystal deposition disease (CPPD), or other autoimmune diseases
* Has any planned surgeries in the upper limbs during the study or any other surgery during the study that would require use of a restricted medication
* Has surgical hardware or other foreign body present in the index shoulder
* Has received an IA corticosteroid of any joint within 3 months of the Screening Visit
* Has received an IA treatment of the index shoulder with any of the following agents within 6 months of the Screening Visit
* Has received intravenous (IV), intrabursal, intratendinous, intramuscular (IM) or epidural corticosteroids within 3 months of the Screening Visit
* Has received oral corticosteroids within 1 month of the Screening Visit
* Has received inhaled, intranasal, or topical corticosteroids within 2 weeks of the Screening Visit
* Has had significant changes to lifestyle with regard to physical activity and lifestyle within 1 month of the Screening Visit or any planned changes throughout the duration of the study
* Has known hypersensitivity to TA or PLGA
* Has laboratory evidence of infection with (HIV), a positive test for hepatitis B surface antigen (HBsAg), or positive serology for hepatitis C virus (HCV) with positive test for HCV ribonucleic acid
* Has an electrocardiogram (ECG) abnormality
* Has uncontrolled diabetes as indicated by a hemoglobin A1c of >8% (>59 mmol/mol).
* Has a history of sarcoidosis or amyloidosis
* Has a history of or active Cushing's syndrome
* Has used chemotherapeutic agents, immunomodulators, or immunosuppressants within 5 years of the Screening Visit
* Has current or history of malignancy within 5 years prior to the Screening Visit, except for basal or squamous cell carcinoma of the skin or cervical carcinoma in situ that has been treated successfully.
* Has active substance use disorder or history of substance use disorder within 12 months prior to the Screening Visit
* Has received a live or live attenuated vaccine within 3 months of the Screening Visit
* Has used any other investigational drug, biologic, or device within 3 months of the Screening Visit
* Has any infection requiring IV antibiotics 4 weeks prior to Day 1 or oral antibiotics 2 weeks prior to Day 1
* Has a contraindication to the use of acetaminophen
* Is a female that is pregnant or nursing or plans to become pregnant during the study; or is a male who plans to inseminate a partner or donate sperm during the study

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (27):
- United States (27):
  - Central Research Associates, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Affinity Orthopedic Specialists, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - TriWest Research Associates, El Cajon, California
  - CORE Orthopedic Medical Center, Encinitas, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Mountain View Clinical Research Center, Denver, Colorado
  - Coastal Orthopaedics and Sports Medicine, Bradenton, Florida
  - South Lake Pain Institute, Clermont, Florida
  - Universal Axon Clinical Research, Homestead, Florida
  - Precision Clinical Research, Lauderdale Lakes, Florida
  - Infinite Clinical Research, Miami, Florida
  - Jewitt Orthopedic Center, Orlando, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Arthritis and Rheumatism Associates PC, Wheaton, Maryland
  - Hassman Research Institute, Berlin, New Jersey
  - M3 Emerging Medical Research, Durham, North Carolina
  - University Orthopedics Center, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Texas Orthopedic Specialists, Bedford, Texas
  - Centex Studies, Inc., Houston, Texas
  - Spectrum Medical, Inc., Danville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population
Started | 7 | 3 | 5 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 3 | 5 | 4
Not completed — Terminated by Sponsor | 7 | 3 | 5 | 2
Not completed — Noncompliance | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population | Total
Number analyzed (Participants) | 7 | 3 | 5 | 4 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The two populations were analyzed separately
  years
    OA Population: number analyzed (Participants) | 7 | 3 | 0 | 0 | 10
    OA Population | 61.7 (13.07) | 60.0 (2.65) |  |  | 61.2 (10.78)
    Adhesive Capsulitis Population: number analyzed (Participants) | 0 | 0 | 5 | 4 | 9
    Adhesive Capsulitis Population |  |  | 56.2 (12.64) | 58.5 (4.80) | 57.2 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The two populations were analyzed separately
  Participants
    OA Population: number analyzed (Participants) | 7 | 3 | 0 | 0 | 10
    OA Population: Female | 1 | 1 |  |  | 2
    OA Population: Male | 6 | 2 |  |  | 8
    Adhesive Capsulitis Population: number analyzed (Participants) | 0 | 0 | 5 | 4 | 9
    Adhesive Capsulitis Population: Female |  |  | 4 | 3 | 7
    Adhesive Capsulitis Population: Male |  |  | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The two populations were analyzed separately
  Participants
    OA Population: number analyzed (Participants) | 7 | 3 | 0 | 0 | 10
    OA Population: Hispanic or Latino | 1 | 0 |  |  | 1
    OA Population: Not Hispanic or Latino | 6 | 3 |  |  | 9
    OA Population: Unknown or Not Reported | 0 | 0 |  |  | 0
    Adhesive Capsulitis Population: number analyzed (Participants) | 0 | 0 | 5 | 4 | 9
    Adhesive Capsulitis Population: Hispanic or Latino |  |  | 1 | 0 | 1
    Adhesive Capsulitis Population: Not Hispanic or Latino |  |  | 4 | 4 | 8
    Adhesive Capsulitis Population: Unknown or Not Reported |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The two populations were analyzed separately
  Participants
    OA Population: number analyzed (Participants) | 7 | 3 | 0 | 0 | 10
    OA Population: American Indian or Alaska Native | 0 | 0 |  |  | 0
    OA Population: Asian | 0 | 0 |  |  | 0
    OA Population: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    OA Population: Black or African American | 1 | 1 |  |  | 2
    OA Population: White | 6 | 1 |  |  | 7
    OA Population: More than one race | 0 | 0 |  |  | 0
    OA Population: Unknown or Not Reported | 0 | 1 |  |  | 1
    Adhesive Capsulitis Population: number analyzed (Participants) | 0 | 0 | 5 | 4 | 9
    Adhesive Capsulitis Population: American Indian or Alaska Native |  |  | 0 | 0 | 0
    Adhesive Capsulitis Population: Asian |  |  | 0 | 0 | 0
    Adhesive Capsulitis Population: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    Adhesive Capsulitis Population: Black or African American |  |  | 1 | 0 | 1
    Adhesive Capsulitis Population: White |  |  | 4 | 4 | 8
    Adhesive Capsulitis Population: More than one race |  |  | 0 | 0 | 0
    Adhesive Capsulitis Population: Unknown or Not Reported |  |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 5 | 4 | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The two populations were analyzed separately
  kg/m^2
    OA Population: number analyzed (Participants) | 7 | 3 | 0 | 0 | 10
    OA Population | 28.95 (2.473) | 30.61 (3.744) |  |  | 29.45 (2.799)
    Adhesive Capsulitis Population: number analyzed (Participants) | 0 | 0 | 5 | 4 | 9
    Adhesive Capsulitis Population |  |  | 33.03 (4.425) | 27.99 (6.752) | 30.79 (5.826)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of the Change From Baseline in the Weekly Mean of the Daily Shoulder Pain With Movement
Description: The pain intensity score is measured using an 11-point numeric rating scale (NRS), where 0 indicates "No pain" and 10 indicates "Worst possible pain."
Time Frame: Baseline to 8 weeks
Population: Due to the early termination of the study, this endpoint was not analyzed. Change from baseline in the weekly mean of the average daily shoulder pain with movement score is included in Outcome Measure 2
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in the Weekly Mean of the Average Daily Shoulder Pain With Movement Score
Description: as for outcome 1
Time Frame: Baseline to 12 weeks
Population: All patients who received a dose of study drug assigned to the FX006 32 mg and the Placebo arm were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population
Number analyzed (Participants) | 7 | 2 | 5 | 2
score on a scale | -3.54 (2.477) | -0.88 (1.237) | -4.05 (2.648) | -1.58 (2.003)

3. Secondary Outcome: Change From Baseline in the SPADI Pain Subscale at Week 12
Description: Shoulder Pain and Disability Index (SPADI) Pain scale is measured using 5 11-point NRS questions where 0 indicates "no pain" and 10 indicates "worst pain imaginable." The Pain and Disability Subscales are presented as a percentage of the total possible score. The Total SPADI score ranges from 0 (best) to 100 (worst) is computed by taking the means of the Pain and Disability Subscale scores.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population
Number analyzed (Participants) | 7 | 3 | 4 | 2
score on a scale | -32.00 (21.385) | -9.33 (26.633) | -52.00 (49.585) | -40.00 (5.657)

4. Secondary Outcome: Change From Baseline in the SPADI Disability Subscale at Week 12
Description: Shoulder Pain and Disability Index (SPADI) Disability scale is measured using 8 11-point NRS questions where 0 indicates "no difficulty" and 10 indicates "so difficult it requires help." The Pain and Disability Subscales are presented as a percentage of the total possible score. The Total SPADI score ranges from 0 (best) to 100 (worst) is computed by taking the means of the Pain and Disability Subscale scores.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population
Number analyzed (Participants) | 6 | 3 | 4 | 2
score on a scale | -32.29 (9.435) | -10.42 (17.559) | -50.94 (31.842) | -50.00 (21.213)

5. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at Week 12
Description: PGIC is measured using a 7-point NRS where 1 indicates "very much improved" and 7 indicates "very much worse."
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population
Number analyzed (Participants) | 6 | 3 | 4 | 2
score on a scale | 2.7 (1.51) | 3.3 (1.15) | 1.5 (0.58) | 2.5 (0.71)

6. Secondary Outcome: Change From Baseline in the Range of Motion (ROM) of Active External Rotation at Week 12
Description: Measured using a goniometer which is a device that measures ROM joint angles
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population
Number analyzed (Participants) | 5 | 3 | 4 | 1
Degrees | -4.76 (13.068) | 7.87 (26.307) | 68.70 (81.850) | -4.60 (NA) — There was only participant analyzed.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until the end of patient participation in the study up to 24 weeks.
Arm/Group | FX006 32mg in Glenohumeral OA Population | Normal Saline in Glenohumeral OA Population | FX006 32mg in Adhesive Capsulitis Population | Normal Saline in Adhesive Capsulitis Population
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 1/7 | 0/3 | 2/5 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32mg in Glenohumeral OA Population (N=7) | Normal Saline in Glenohumeral OA Population (N=3) | FX006 32mg in Adhesive Capsulitis Population (N=5) | Normal Saline in Adhesive Capsulitis Population (N=4)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor due to the COVID-19 pandemic. Summary statistics were calculated for available data, but given that only approximately 8% of the planned study population had enrolled and there no conclusions can be drawn from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT04160091/Prot_SAP_002.pdf